CLINICAL TRIAL: NCT03971760
Title: Ideal Drainage Output of Post-operative Neck Suction Drain: a Randomized Controlled Trial
Brief Title: Ideal Drainage Output of Post-operative Neck Suction Drain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID pandemic
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18.300
Record Dates: First submitted 2019-05-22; First posted 2019-06-03 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Head and Neck Neoplasms; Drain Site Complication; Neck Dissection
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: 30cc/24h (Active Comparator): This group represents the currently used value of drain output used to determine the timing of drain removal
  Interventions: Other: Suction drain removal
- Group 2: 50cc/24h (Experimental): This group represents the experimental value of drain output used to determine the timing of drain removal
  Interventions: Other: Suction drain removal

INTERVENTIONS:
Other: Suction drain removal — Removal of negative pressure suction drain left in place to drain the surgical space after a neck surgery

SUMMARY:
A precautionary measure that is frequently used after a neck surgery is the usage of suction drains, which allow the evacuation or air and fluids accumulated at the site of the surgery using negative pressure. Theoretically this helps promote better healing of the wound. Usage of suction drains, however, requires keeping some patients hospitalized after surgery for drain surveillance while they could have otherwise been discharged to safely begin their convalescence at home. In other cases, patient hospitalisation can be prolonged by the usage of suction drains, because surgeons wait for the output of the drain to fall below a certain quantity before removing them. This of course results in additional costs to the health system. The quantity below which the drain output should fall before drain removal is however not something agreed upon in the medical literature and is generally based on a surgeon's personal experience or that of the institution in which they practice. It would be important to better define this value, since prolonged usage of suction drains is not risk-free. Indeed, they constitute, among other things, an access for bacteria to cause an infection to develop inside the neck, which compromises wound healing and may result in more pronounced scarring. This study aims to compare a frequently used output value (30 mL per 24 hours) with a more permissive one of 50 mL per 24 hours. The investigators will look more specifically at wound complications, length of hospitalisation and cost-effectiveness for the health system. This study will recruit patients undergoing neck surgery at the Centre Hospitalier de l'Université de Montréal to compare both of these suction drain output values.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older of age
* Patient having undergone neck surgery at the CHUM
* Patient operated by an Ear Nose and Throat - Head and Neck surgeon at the CHUM
* Patient with at least one suction drain left post-operatively

Exclusion Criteria:

* Non-suction drain (e.g. capillarity)
* Free-flap reconstruction cases
* Patient with past surgical history of neck dissection
* Patient with pas medical history of radiation therapy in the head and neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Duration of drainage | At the time of patient discharge from the ward, usually up to 1 week
  The length of time during which the suction drain is left in place, from the time of the surgery to the time of drain removal

SECONDARY OUTCOMES:
Seroma rate | Up to 6 weeks following surgery
  The rate of seroma as wound complication, defined as an accumulation of serous fluid in the surgical space

OTHER OUTCOMES:
Duration of admission | At the time of patient discharge from the ward, usually up to 1 week
  Length of patient's stay in hospital after surgery
Wound infection | Up to 6 weeks following surgery
  Surgical site infection following surgery